CLINICAL TRIAL: NCT03492736
Title: Does Melatonin Improve Neurocognitive Function, Cardiovascular Outcomes and Control of Breathing in Untreated Obstructive Sleep Apnea?
Brief Title: Effects of Melatonin in Untreated Obstructive Sleep Apnea
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI leaving the laboratory
Sponsor: Naomi Deacon (Other)
Responsible Party: Sponsor-Investigator, Naomi Deacon, Research Scholar, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 180013
Record Dates: First submitted 2018-04-02; First posted 2018-04-10 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Experimental): 30 days 10mg Melatonin taken nightly 1 hour before bed
  Interventions: Dietary Supplement: Melatonin
- Placebo (Placebo Comparator): 30 days placebo taken nightly 1 hour before bed
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Melatonin — 30 days 10mg Melatonin taken nightly 1 hour before bed
  Arms: Melatonin
Other: Placebo — 30 days placebo taken nightly 1 hour before bed
  Arms: Placebo

SUMMARY:
The investigators have previously shown that 1 week of 10mg Melatonin improves sleep consolidation in untreated obstructive sleep apnea (OSA) patients. This study aims to extend on those findings to determine if longer treatment of Melatonin improves other outcomes in untreated OSA patients.

DETAILED DESCRIPTION:
Intermittent hypoxia (low oxygen), sleep fragmentation and restriction are characteristic of obstructive sleep apnea (OSA) and cause mental deficits and cardiovascular disease (CVD). Melatonin (MLT) is a hormone with sleep promoting properties and the investigators have found 7 days 10mg MLT treatment significantly increases sleep consolidation in untreated OSA. Thus, melatonin could improve mental function. MLT also has potent antioxidant, anti-inflammatory and anti-hypertensive properties. In humans with CVD and metabolic disorder exogenous MLT improves a wide range of cardio-metabolic outcomes. In rat models of OSA, MLT completely blocks intermittent hypoxia induced cardiovascular damage and brain cell death. Intermittent hypoxia also induces lasting changes in the neural control of breathing, which worsens OSA. Experimentally antioxidants block the induction of changes to neural control of breathing. Thus MLT may also normalize the control of breathing and reduce the severity of OSA. Given these findings, the hypothesis is that MLT will improve mental function, cardiovascular outcomes and control of breathing in untreated OSA.

ELIGIBILITY:
Inclusion Criteria:

* moderate-severe OSA (AHI ≥15/hr)

Exclusion Criteria:

* non-English speakers (due to necessity to complete neurocognitive testing)
* other sleep disorders
* history of driving or other accidents due to sleepiness or an Epworth score (ESS)> 18
* pregnant
* smokers (quit ≥ 1 year ago acceptable)
* diabetes
* cardiac (other than hypertension), pulmonary, renal, neurologic, neuromuscular or hepatic disease
* Substantial alcohol (>3oz/day) or use of illicit drugs
* psychiatric disorders (other than depression or anxiety)
* current MLT use or use within last 6 months
* beta blockers, central nervous system depressants or stimulants, anti-inflammatories, anticoagulants, immunosuppressants, vitamins, antioxidants.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Groups will be matched for gender, age and BMI
Enrollment: 1 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
PHQ-9 score | baseline versus on the 30th day of treatment
  9 Questions relating to depressive symptoms. Answers to each question rank from 0-3. Minimum total score = 0, maximum total score = 27, with >=10 indicating clinically significant moderate severity depressive symptoms.

SECONDARY OUTCOMES:
Reactive Hyperemia Index | baseline versus on the 30th day of treatment
  Endothelial function is calculated as the ratio between the magnitude of the mean post-occlusion pulse wave amplitude and mean baseline pulse wave amplitude.

OTHER OUTCOMES:
Hypoxic ventilatory response | baseline versus on the 30th day of treatment
  change in ventilation per change in expiratory CO2 during sustained hypoxia

CONTACTS AND LOCATIONS:
Overall Officials: Naomi L Deacon, Ph.D., Study Director — UCSD Pulmonary and Sleep Medicine
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No